CLINICAL TRIAL: NCT01798927
Title: Investigation of Lower Extremity Orthoses on Gait in Persons With Parkinson's Disease: a Case Series.
Brief Title: Effect of Lower Extremity Ankle Foot Orthoses in Parkinson's Disease
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Modifications are being made to protocol
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Karen McCain, Assistant Professor, University of Texas Southwestern Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PD AFO
Record Dates: First submitted 2013-02-11; First posted 2013-02-26 (Estimated); Results first posted 2015-08-03 (Estimated); Last update posted 2015-08-03 (Estimated); Status verified 2015-07

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's disease; ankle foot orthosis (AFO); gait
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ankle foot orthosis fitting (Other): All participants will receive ankle foot orthosis or orthoses. Outcomes will be compared to pre-bracing findings.
  Interventions: Device: Ankle foot orthosis

INTERVENTIONS:
Device: Ankle foot orthosis — Participants will receive a Tamarack ankle foot orthosis with a check strap for gait training as well as a home walking program.
  Other Names: Tamarack with check strap

SUMMARY:
The purpose of this study is to investigate the impact of a specifically designed ankle foot orthosis (AFO, hinged, with Tamarack joint and adjustable check strap) on the spatial and temporal gait parameters, electromyography (EMG) and walking endurance, in select individuals living with Parkinson's disease.

DETAILED DESCRIPTION:
This study will be 10 weeks long. Following fitting with unilateral or bilateral custom-fabricated AFOs the subject will participate in 4 gait training sessions which will be at weeks 1, 2, and 7. Each training session will be 45-60 minutes in duration. Various outcome measures will be completed at the following times: time of consent (T1), treatment 1 at time of brace delivery (T2), week 5 (T3), and week 10 (T4). Subjects will be closely monitored throughout the 10 week study and will be unenrolled by self-request or the following medical reasons: 1. New diagnosis with direct consequences affecting gait training, 2. Inability to tolerate the study AFO(s).

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of Parkinson's Disease
* Between the ages of 50 and 75
* Ability to walk 150 feet independently over level surfaces with or without an assistive device
* Stable medication usage for the duration of the study (10 weeks)
* Obvious gait dysfunction (Observational Gait Analysis)
* Score of greater than 22 on the Short Orientation-Memory-Concentration Test

Exclusion Criteria:

* Body mass index of greater than 35
* Dorsiflexion range of motion less than neutral (90 degrees)
* Any other uncontrolled health condition for which gait training is contraindicated

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2012-12; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karen J McCain, DPT, Principal Investigator — UTSW Medical Center
Locations (1):
- UT Southwestern Medical Center, School of Health Professions, Dallas, Texas, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ankle Foot Orthosis Fitting
Started | 4
Completed | 3
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Ankle Foot Orthosis Fitting
Number analyzed (Participants) | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 68 (5.22)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 4
Region of Enrollment [Number; unit: participants]
  United States | 4

OUTCOME MEASURES:

1. Primary Outcome: Change in Step Length by Means of Computerized Gait Analysis From Initial to Final Testing
Description: Participants will be asked to walk on a 12-16 foot long vinyl pad placed on the floor. The mat will record and analyze step length.
Time Frame: Done at time of enrollment in the study, i.e. baseline and 10 weeks post enrollment
Population: step length was analyzed from the GAITRite
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Ankle Foot Orthosis Fitting
Number analyzed (Participants) | 3
cm | 6.7 (2.77)

2. Secondary Outcome: Number of Participants With a Change in Electromyography of Key Lower Extremity Muscles From Initial to Final Testing
Description: Surface electromyography will be done on key muscles in the lower extremity (quads, anterior tibialis, gastrocnemius) during computerized gait assessment. Changes in EMG activity include things such as increases in amplitude or timing that might indicate increases in strength or motor learning as a result of wearing the ankle foot orthosis.
Time Frame: Done at time of enrollment in the study, i.e. baseline and week 10 post enrollment.
Population: EMG data was analyzed from 3 of the 4 participants
Measure: Number; unit: participants
Arm/Group | Ankle Foot Orthosis Fitting
Number analyzed (Participants) | 3
participants | 0

3. Other Pre Specified Outcome: Change in Walking Endurance by Use of 6-Minute Walk Test From Initial to Final Testing
Description: Each participant will be asked to walk at a self-selected velocity on level surfaces for 6 minutes. They will be allowed to use assistive devices if necessary.
Time Frame: Done at time of enrollment in the study, i.e. baseline and week 10 post enrollment
Population: data from 3 of the 4 participants was analyzed
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Ankle Foot Orthosis Fitting
Number analyzed (Participants) | 3
meters | .2 (0)

ADVERSE EVENTS:
Arm/Group | Ankle Foot Orthosis Fitting
Serious Adverse Events (participants affected / at risk) | 0/3
Other Adverse Events (participants affected / at risk) | 0/3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No